CLINICAL TRIAL: NCT03666182
Title: The Relationship Between Genetics, Body Mass Index, Fat Intake, Fat Taste Sensitivity and Food Preference
Brief Title: Genetics and Fat Taste Sensitivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2017-18_138
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Taste Sensitivity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole Sample: Female, Caucasian participants aged 18-65 years.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
A cross-sectional quantitative study will be carried out; recruiting female, Caucasian participants aged 18-65 years. The relevance of candidate gene studies is disputed. Research has shown associations between genotype and total fat intake. However, food preference is often described as a result of exposure to food types during upbringing. Many single nucleotide polymorphisms (SNP) have been associated with fat taste sensitivity, the majority of research shows that with a reduced sensitivity comes a higher total fat consumption.

This study aims to assess the relationship between rs1761667 genotype, body mass index, fat intake, fat taste sensitivity and fat taste preference.

ELIGIBILITY:
Inclusion Criteria:

* European Citizen.
* Caucasian
* Aged between 18-65 years.
* Female

Exclusion Criteria:

* Currently following a diet or weight loss plan or have not been for over 6 months of the previous year.
* Suffering from diabetes (type I or II).
* Have cancer, or have not had cancer in the past.
* Smoker.
* Pregnant.
* Lactose intolerant .

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: European Citizen, Caucasian, Aged between 18-65 years, Female
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-11 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | September - November 2018

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No